CLINICAL TRIAL: NCT06439160
Title: Exploring the Changes in Social Interaction and Its Protective Features in Anorexia Nervosa
Acronym: SOCINTERACAN
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: University of Turin, Italy (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Other Study IDs: 49C401
Record Dates: First submitted 2024-05-20; First posted 2024-06-03 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Social interaction; Rehabilitation
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- anorexia nervosa/AN: Individuals of both biological sexes affected by AN who will take part in the multidisciplinary inpatient intensive rehabilitation treatment as offered by the U.O. dei Disturbi del Comportamento Alimentare, San Giuseppe Hospital, Piancavallo (VCO), Italy.
  Inclusion Criteria:
  i) age between 18 and 65 years old; ii) diagnosis of AN, as per DSM V criteria (APA, 2013); iii) BMI ≤ 17 Kg/m2; iv) adherence to the rehabilitation program, meaning participating at the 75% of the proposed activities.
  Exclusion criteria:
  i) presence of other pathologies not associated with AN (i.e., neurodegenerative diseases); ii) severe psychopathologies other than AN (i.e., schizophrenia); iii) spontaneous dropout from the multidisciplinary inpatient intensive rehabilitation treatment.
  Interventions: Other: Participants will be asked to complete a series of questionnaires at t0, t1 and t2

INTERVENTIONS:
Other: Participants will be asked to complete a series of questionnaires at t0, t1 and t2 — Individuals will be people who voluntarily will take part in a residential three to six weeks multidisciplinary inpatient intensive rehabilitation treatment targeting the improvement of psychological well-being, body image, and psychopathology for anorexia nervosa.
  Therefore, at T0 (at the beginning of the treatment) and T1 (at the end of the rehabilitation programme), participants will fill out some self-report questionnaires to evaluate the effect of the multidisciplinary inpatient intensive rehabilitation treatment on different outcomes (i.e. psychological well-being, eating pathology, body image, and comorbidities), among which their social components/skills. Moreover, we will ask participants to complete 3 months after discharge the questionnaires related to the social components/skills only. Participants will be contacted by email, within the email participants will find a link to click on for the completion of the questionnaires.

SUMMARY:
Anorexia Nervosa (AN) is an eating disorder often characterised by restriction of food intake, being underweight, body image uneasiness, and the possibility of binge eating, purging, fasting behaviours, and excessive exercising. Despite weight and eating habits being one, and perhaps the most recognizable, components of AN, AN is a multidimensional disease. For example, individuals affected by AN might show psychological suffering, such as depression and anxiety. For example, social anxiety disorder/social phobia is the first or second most common comorbid anxiety in AN (i.e. prevalence rates ranging from 16% to 88.2% in AN against 12% in the general population). Moreover, the highest the level of social anxiety the highest the severity of the eating disorder psychopathology. This latter component resonates with findings on the difficulties observed in people affected by AN in creating and maintaining satisfactory relationships with others. These evidences tell us the importance to take into account the social components/skills of people affected by AN.

The development of social components/skills of people affected by AN during their recovery can be considered as a protective factor for future relapse. This would be of relevance for the creation of rehabilitative programs.

DETAILED DESCRIPTION:
Anorexia Nervosa (AN) is an eating disorder often characterised by restriction of food intake, being underweight, body image uneasiness, and the possibility of binge eating, purging, fasting behaviours, and excessive exercising. AN is of relevance for the health care system because of the high mortality rates, high psychiatric comorbidity, high suicide risk, and because of the high costs for the health system. Despite weight and eating habits being one, and perhaps the most recognizable, components of AN, AN is a multidimensional disease. For example, individuals affected by AN might show psychological suffering, such as depression and anxiety. For example, social anxiety disorder/social phobia is the first or second most common comorbid anxiety in AN (i.e. prevalence rates ranging from 16% to 88.2% in AN against 12% in the general population). Moreover, the highest the level of social anxiety the highest the severity of the eating disorder psychopathology. This latter component resonates with findings on the difficulties observed in people affected by AN in creating and maintaining satisfactory relationships with others. These evidences tell us the importance to take into account the social components/skills of people affected by AN. Therefore, we believe it would be relevant to understand whether our treatments change the social components/skills of the people affected by AN who access our ward's multidisciplinary inpatient intensive rehabilitation treatment. Moreover, it would be important to evaluate the protective role of participants' social components/skills in the changes in their psychopathology. Despite our rehabilitative activities not having a specific focus on sociality, the activities are conducted on a 1:1 or group basis. This means that our activities have an intrinsic relational and socializing value.

The purpose of the study lays on two outcomes:

* Primary outcome: evaluation of the short-term effects (T0 vs T1) of the multidisciplinary inpatient intensive rehabilitation treatment on the social components/skills of people affected by AN.
* Secondary outcome: evaluation of the long-term effects (T0 vs T2) of the multidisciplinary inpatient intensive rehabilitation treatment on the social components/skills of people affected by AN.

The development of social components/skills of people affected by AN during their recovery can be considered as a protective factor for future relapse. This would be of relevance for the creation of rehabilitative programs

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years old;
* diagnosis of AN, as per DSM V criteria (APA, 2013);
* BMI ≤ 17 Kg/m2;
* adherence to the rehabilitation program, meaning participating at the 75% of the proposed activities.

Exclusion criteria:

* presence of other pathologies not associated with AN (i.e., neurodegenerative diseases);
* severe psychopathologies other than AN (i.e., schizophrenia);
* spontaneous dropout from the multidisciplinary inpatient intensive rehabilitation treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals of both biological sexes affected by AN who will take part in the multidisciplinary inpatient intensive rehabilitation treatment as offered by the U.O. dei Disturbi del Comportamento Alimentare, San Giuseppe Hospital, Piancavallo (VCO), Italy.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) | Through study completion, an average of 4 months
  Social anhedonia will be evaluated by the Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS). This self-report questionnaire is made up of 17-item for measuring individuals' tendency to look forward to interactions with others (anticipatory interpersonal pleasure - 7 items) and the experienced pleasure in social interactions (consummatory interpersonal pleasure - 10 items). The ACIPS is scored on a six-point Likert scale ranging from 1 (very false for me) to 6 (very true for me).
The Social Appearance Anxiety Scale (SAAS) | Through study completion, an average of 4 months
  The scale will be used to assess anxiety about being negatively evaluated by others because of one's overall appearance, including body shape (e.g., "I am concerned people would not like me because of the way I look and I am afraid that people find me unattractive"). The scale contains 16 items rated on a 5-points Likert scale ranging from 1 = not at all to 5 = extremely, with higher scores reflecting a higher social appearance anxiety scale.
The Social Interaction Anxiety Scale (SIAS) | Through study completion, an average of 4 months
  The scale will be used to assess the fear of interacting in dyads and groups (e.g., ''I have difficulty talking with other people''). The scale contains 20 items rated on a 5-points Likert scale ranging from 0 = not at all to 4 = extremely, with a higher score indicating greater social interaction anxiety
Social Phobia Scale (SPS) | Through study completion, an average of 4 months
  We will administer the scale to evaluate the fear of being scrutinized by others during routine activities, such as eating, drinking, or writing (e.g., ''I become anxious if I have to write in front of other people''). The scale is made up of 20 items rated on a five-points Likert scale ranging from 0 = not at all to 4 = extremely, with a higher score indicating greater fear of scrutiny.

CONTACTS AND LOCATIONS:
Locations (1):
- istituto Auxologico italiano IRCSS, Milan, MI, Italy